CLINICAL TRIAL: NCT04580667
Title: Prospective Observational Exploratory Clinical Study to Determine the Assay Cut-Off for the RadTox Test in Prostate Cancer Patients to Predict Gastrointestinal Radiation Toxicity Using Circulating Cell Free DNA Directly From Plasma
Brief Title: Determination of Assay Cut-Off for the RadTox Test in Prostate Cancer Patients to Predict GI Radiation Toxicity
Status: Withdrawn | Type: Observational
Why Stopped: The sponsor declared bankruptcy
Sponsor: DiaCarta, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DIA.0009
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Evaluate toxicity biomarkers: Investigators will determine if measurement of circulating DNA from normal tissues shortly after the start of radiotherapy provides an early indication of patients at high risk of radiation-related toxicity. Blood specimens for RadTox test will be collected: (a) prior to radiotherapy (T0); (b) after the 2nd but before the 4th radiotherapy dose during week 1 (T1); (c) on Week 2 during radiotherapy (T2); and (d) 3 months after completion of radiotherapy (T3).
  Interventions: Other: Collection of plasma samples

INTERVENTIONS:
Other: Collection of plasma samples — Collection of plasma samples - Plasma samples are collected at different times during the study for the RadTox test.

SUMMARY:
This clinical study is conducted to develop a new test to identify prostate cancer patients at highest risk of radiotherapy-related complications, especially related to gastrolintestinal (GI) toxicities. This clinical study would allow monitoring of total tissue damage in blood samples as early as after the 2nd but before the 4th radiotherapy dose during week 1 of radiotherapy, which could help clinicians make treatment decisions. Detection of excessive tissue damage at this early time, well before symptoms occur, could allow doctors to tailor interventions which could include patient therapies that would reduce or prevent the problems that occur due to radiotherapy of their cancer.

DETAILED DESCRIPTION:
Currently, a patient's risk for toxicity is based almost exclusively on population statistics. Radiation (and chemotherapy) doses are based on phase I data and not on the individual's specific genetics or hidden predispositions. RadTox measures cell damage as early as after the 2nd but before the 4th radiotherapy dose during week 1 of radiotherapy and should help identify patients at high risk for radiation complications. This should allow physicians to adjust radiation field size and dose to minimize long-term toxicity, especially gastrointestinal toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with adenocarcinoma of the prostate who have not received previous treatment (defined as prostatectomy, transurethral resection of the prostate [TURP], radiation of the pelvis, and GreenLight Laser Therapy) except for short-term (≤6 months) Androgen Deprivation Therapy (ADT) according to National Comprehensive Cancer Network (NCCN) guidelines.
* Candidate for definitive prostate radiotherapy (either IMRT or proton).
* Patients to be treated with IMRT should have all radiation treatment planned with IMRT, whereas patients to be treated with protons should have all radiation treatment planned with protons (including pelvic nodes if treated).
* Localized prostate cancer, as confirmed by staging with Prostate-Specific Antigen (PSA), biopsy, Gleason score, and clinical stage.
* Nuclear medicine bone imaging is required for confirmation of the absence of overt metastatic disease in bones if any high-risk criteria are identified (clinical stage T3a or higher; or 1-4 cores of Gleason score 8 [NCCN Grade Group 4] or 4+5; or PSA ≥20 ng/mL).
* Diagnosed with any of the NCCN initial groups (i.e., Very-Low-Risk, Low-Risk, Intermediate-Risk [both Favorable and Non-Favorable Intermediate-Risk]; High-Risk; or Very-High-Risk) (see Appendix III for NCCN classifications of various risk groups). For Very-High-Risk, subjects are to have negative prostate cancer specific PET/CT imaging for confirmation of being metastasis free.
* The score for Question 16 (i.e., "Overall, how big a problem have your bowel habits been for you during the last 4 weeks?") of the Bowel Habits section of Expanded Prostate Cancer Index Composite (EPIC) questionnaire must be 2 or below.
* 30-85 years of age at the time of consent.
* Eastern Cooperative Oncology Group (ECOG)/Zubrod Performance Status 0 - 2.

Exclusion Criteria:

* Findings of metastatic disease (nodal or distant, >N1 or M1).
* Prior prostatectomy, TURP, radiation of the pelvis, or GreenLight Laser Therapy.
* History of invasive rectal malignancy or other pelvic malignancy, regardless of disease-free interval.
* The score for Question 16 (i.e., "Overall, how big a problem have your bowel habits been for you during the last 4 weeks?") of EPIC questionnaire is 3 or above.
* Active inflammatory bowel disease (i.e., patients requiring medical interventions or who are symptomatic) or documented history of inflammatory bowel disease requiring intervention.
* Prior pelvic radiotherapy for any reason.
* Documented lack of psychological ability or general health permitting completion of the study requirements and required follow-up.
* Documented decisionally impaired persons who have a diminished capacity to understand the risks and benefits of participation in research and to autonomously provide informed consent.
* Subjects who participated in a clinical trial of an investigational device, drug or biologics within the past 30 days.
* Subjects who are currently undergoing any cancer drug treatment. However, patients who had received cancer drug treatment and stopped the treatment for >4 weeks prior to the start of radiotherapy can be included. (Hormone therapy is allowed if judged appropriate and necessary by the treating physicians.)

Ages: 30 Years to 85 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on the presence of prostate cancer.
Study Population: Male patients with undergoing radiation therapy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
To determine the cut-off values from the RadTox test results during early radiation treatment from all evaluable subjects to differentiate high toxicity score from average or low toxicity score. | 1 year after radiotherapy
  The cut-off values of all evaluable subjects will be measured based on the Receiver Operating Characteristic (ROC) analysis to optimize detection of true high-risk patients with ≥60% sensitivity and ≥60% specificity allowing for an acceptable number of high-risk classified but normal-risk patients.

SECONDARY OUTCOMES:
To determine the cut-off values from the RadTox test performed during early radiation treatment with patients categorized according to demographics and treatment options to differentiate high toxicity score from average or low toxicity score. | 1 year after radiotherapy
  The RadTox test results will be measured to determine the cut-off values according of patients' demographics and treatment options such as fractionation and radiation modality.

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Vallerga, PhD, MBA, Principal Investigator — DiaCarta, Inc.
Locations (5):
- United States (5):
  - University of Florida, Gainesville, FL, Gainesville, Florida
  - UF Health Proton Therapy Institute, Jacksonville, Florida
  - NY Cancer and Blood Specialists, New York, New York
  - NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - NY Cancer and Blood Specialists, The Bronx, New York